CLINICAL TRIAL: NCT00710086
Title: Remifentanil Intravenous Patient-controlled Labor Analgesia for Nulliparous Women
Brief Title: Intravenous Remifentanil for Labor Analgesia
Acronym: IRELAN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Collaborators: HRSA/Maternal and Child Health Bureau (U.S. Federal Agency)
Responsible Party: XiaoFeng Shen, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NJFY-08021MZ; NSR083
Record Dates: First submitted 2008-07-02; First posted 2008-07-04 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Labor Pain
Keywords: Remifentanil; Patient-controlled analgesia; Intravenous analgesia
MeSH Terms: conditions — Labor Pain | interventions — Hydromorphone; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Intravenous administration of hydromorphone intermittently
  Interventions: Drug: Hydromorphone
- 2 (Experimental): Remifentanil intravenous patient-controlled analgesia
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Hydromorphone — Intravenous administration of hydromorphone 1mg at the patient's request if they felt uterine contraction pain
  Arms: 1
Drug: Remifentanil — Remifentanil intravenous PCA: 0.2μg/kg, lockout time interval 2 minutes, continuous infusion rate 0.2-0.8μg/kg/min.
  Other Names: ReiFen
  Arms: 2

SUMMARY:
Labor analgesia is an essential health caring procedure for women. However, epidural analgesia cannot be performed on all subjects for different contraindications, such as lower platelet counter, back infection at the puncture site, and fear of epidural injection etc. Therefore, intravenous analgesia is an alternative for such conditions. Given the influence of intravenous administration of drugs on fetus, the drug selection is very important. Remifentanil, a super-short efficacious opioid, can last for 3-4 minutes after injection, which is similar in both maternal and fetal environment. Thus the fetus-associated side effects would be less than other drugs. The investigators hypothesized that remifentanil would be a superior intravenous drug used with patient-controlled technique for labor analgesia.

ELIGIBILITY:
Inclusion Criteria:

1. Nulliparous women
2. > 18 years and < 45 years
3. Spontaneous labor
4. Analgesia request
5. Epidural puncture contraindications
6. Tendency of bleeding

Exclusion Criteria:

1. Allergy to opioids, a history of the use of centrally-acting drugs of any sort, chronic pain and psychiatric diseases records
2. Participants younger than 18 years or older than 45 years
3. Those who were not willing to or could not finish the whole study at any time
4. Using or used in the past 14 days of the monoamine oxidase inhibitors
5. Alcohol addictive or narcotic dependent patients were excluded for their influence on the analgesic efficacy of the epidural analgesics
6. Subjects with a nonvertex presentation or scheduled induction of labor
7. Cervical dilation was 5.0cm or greater before performing epidural puncture and catheterization
8. Diagnosed diabetes mellitus and pregnancy-induced hypertension
9. Twin gestation and breech presentation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1000 (Actual)
Dates: Start 2008-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Maternal Visual Analog Scale (VAS) rating of pain | Prior to analgesia, latent phrase, active phrase, second stage of labor, posterior to vaginal delivery

SECONDARY OUTCOMES:
Rate of cesarean delivery | Analgesia initiation (0 min) to successful vaginal delivery (this time period underwent changing in different individuals)
Rate of instrument-assisted delivery | Analgesia initiation (0 min) to successful vaginal delivery (this time period underwent changing in different individuals)
Indications of cesarean delivery | Analgesia initiation (0 min) to cesarean section (this time period underwent changing in different individuals)
Duration of analgesia | Initiation of analgesia (0 min) to the disappearance of sensory block (this time period underwent changing in different individuals)
Maternal satisfaction with analgesia | At the end of the vaginal delivery (this time period underwent changing in different individuals)
Maternal oral temperature | Analgesia initiation (0 min) to successful vaginal delivery (this time period underwent changing in different individuals)
Use of oxytocin after analgesia | Analgesia initiation (0 min) to successful vaginal delivery (this time period underwent changing in different individuals)
Maximal oxytocin dose | At the end of vaginal delivery (this time period underwent changing in different individuals)
Breastfeeding success at 6 weeks after vaginal delivery | At the sixth week after successful delivery
Neonatal one-minute Apgar scale | At the first minute of baby was born
Neonatal five-minute Apgar scale | At the fifth minute of baby was born
Umbilical-cord gases analysis | At the time baby was born (0 min)
Neonatal sepsis evaluation | After the baby was born (15 min after delivery)
Neonatal antibiotic treatment | After the baby was born (one day after delivery)
Incidence of maternal side effects | Analgesia initiation (0 min) to successful vaginal delivery (this time period underwent changing in different individuals)

CONTACTS AND LOCATIONS:
Overall Officials: XiaoFeng Shen, MD, Study Director — Nanjing Medical University
Locations (1):
- Nanjing Maternal and Child Health Care Hospital, Nanjing, Jiangsu, China